CLINICAL TRIAL: NCT02968030
Title: Influence of a Strengthening Exercise Program for Lower Limbs in Functional Mobility From Irregularly Active Elderly
Brief Title: Strengthening in Functional Mobility of Active Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lislei Jorge Patrizzi (Other)
Responsible Party: Sponsor-Investigator, Lislei Jorge Patrizzi, Phd, Universidade Federal do Triangulo Mineiro
Organization: Universidade Federal do Triangulo Mineiro (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEP UFTM 1480
Record Dates: First submitted 2016-11-16; First posted 2016-11-18 (Estimated); Last update posted 2016-12-28 (Estimated); Status verified 2016-10

CONDITIONS: Aged; Muscle Strength
Keywords: Aged; Postural balance; Muscle strength
MeSH Terms: interventions — Muscle Strength; Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Muscle strength (Experimental): Evaluate the effects of a eight weeks program of strengthening exercise on balance and functional mobility in irregular active elderly women
  Interventions: Other: Muscle strength

INTERVENTIONS:
Other: Muscle strength — Strength training The strength training for lower limbs muscles occurred twice a week, 40 minutes per session for eight consecutive weeks.
  n the first two weeks of training, each elderly performed the exercises with 50% of its load defined in 8RM test, increasing to 60 and 70% of the load in the third and fourth subsequent weeks, respectively. After this period, a new evaluation by 8RM strength test was conducted, adopting the fifth and sixth weeks of training 50% of value of the new load defined in 8RM test and to finalize the program in seventh and eighth weeks applied, respectively, 60% and 70% of the new charge. The exercises were performed for the quadriceps, hamstrings, muscles adductor and abductor hip.
  Other Names: Resistance Training; Strength Training

SUMMARY:
Aging is characterized by functional losses among which, the related to mobility and balance may be highlighted. Regular physical activity, including muscle strengthening exercises, is beneficial to a healthy elderly. Thus, this study aimed to verify the influence of 8 weeks-program of lower limbs strengthening exercises in the balance and functional mobility of physically active elderly. The investigators evaluated 18 women, with ages between 61 and 80 years. Balance assessment was performed using the Functional Reach Test (FRT), Timed Up and Go (TUG) test and Romberg test in stable or unstable soil. For muscular strengthening of the lower limbs, the workload was determined by the strength reached in the eight-repetition maximum test (8RM), applying progressive load increments between training sessions conducted (50% , 60% , 70% of 8RM), with the muscle strength being reevaluated in the fourth week of training, with subsequent adjustment of the load for the subsequent training. The training took place in two weekly meetings, in 40-minute sessions, during eight weeks. Data were analyzed using the paired-t test and ANOVA with repeated measures. Among 18 evaluated elderly women, 7 completed the 8 week training proposed. Decrease in TUG time (p = 0,035) and statistically significant increase in muscle strength were observed in all muscle groups trained (quadriceps, hamstrings, adductors and abductors). FRT (p = 0.170) was not significantly different after training. Therefore, strength training proposed was efficient in improving muscle strength in the lower limbs of irregular physically active elderly, impacting positively on functional gain gait. However, the gain in muscle strength was not enough to generate significant results in static balance probably due to the type of exercise performed as well as due being limited to muscle groups of the lower limbs.

ELIGIBILITY:
Inclusion Criteria:

* aged between 61 and 80
* irregularly active (IPAQ)

Exclusion Criteria:

* Presence of one or more of the following conditions: neurological diseases, impaired cognitive autonomy or limited self-determination capacity, limiting orthopedic injury, orthoses for lower limb, hip or knee prosthesis, the cardiorespiratory system diseases or any kind of commitment that prevented the permanence in the standing position.

Ages: 61 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2008-01; Primary Completion 2008-07 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Functional mobility | The results were obtained at the end of the eight weeks of intervention
  The TUG allows a quantitative assessment of gait and mobility, enabling the investigation of the effects of a particular intervention on these parameters (Van Iersel et al., 2008). The TUG is a sensitive test, is a good option of choice to be used as the primary outcome measure in clinical trials to improve gait and mobility (Van Iersel et al., 2008). It allows the researcher to observe the sitting balance of transfers from sitting to standing position and vice versa, as well as stability while walking and walking course changes.
  For the application of TUG has asked the elderly up from a chair without armrest from the recumbent position, wander around a distance of 3 meters safely and quickly, turn, return on the same route and the chair again with the back supported on back. Performance was assessed by timing the time required for the completion of the test. The time taken for the test is determining the risk for falls, classified as low, when the time spent on the test is less than
Risk of falls and Balance | The results were obtained at the end of the eight weeks of intervention
  To the risk of falls in the elderly, the Romberg test is an effective method, since its completion provides anteroposterior instability or increased body sway. For this test, in the standing position the participants remained with the feet together, aligned head and arms along the body. Then, it was requested that, keeping the position described, the participants close their eyes for a period of 30 seconds. Later, the same test was repeated, but on shaky ground when the participant was left standing position on a foam surface, requesting again the closing of the eyes. A procedure again observing the imbalance with time record in seconds, before its occurrence.

SECONDARY OUTCOMES:
Muscle strength | The results were obtained at the end of the eight weeks of intervention
  To evaluate muscle strength and determination of the optimal load training to strengthen the lower limbs the investigators used the strength test eight maximum repetitions (8RM) for each proposed exercise. The 8RM test corresponded to the maximum load that could be raised by the participants throughout the normal range of motion, maintaining the proper technique in eight repetitions (Canuto et al., 2011). Before starting the test was performed 8RM heating with 10 repetitions without any charge to the motion that would run the test and after two minutes the test was started. The materials used were shinguards 0.5 kg to 5 kg.

CONTACTS AND LOCATIONS:
Locations (1):
- Lislei Jorge Patrizzi, Uberaba, Minas Gerais, Brazil